CLINICAL TRIAL: NCT06593483
Title: Increasing Effectiveness of an Alcohol Use Reduction Exercise Using Self-Talk Videos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Emily Grekin, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-10-6241
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Heavy Drinking
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Assessment Only (No Intervention)
- Motivational Interview Only (Active Comparator)
  Interventions: Behavioral: Motivational Interviewing
- Motivational Interview Plus Video (Experimental)
  Interventions: Behavioral: Motivational Interview with Self-Talk Video

INTERVENTIONS:
Behavioral: Motivational Interview with Self-Talk Video — Participants will engage in an interview based in motivational interviewing techniques and then record a self talk video discussing their goals and reasons for reducing their drinking.
  Arms: Motivational Interview Plus Video
Behavioral: Motivational Interviewing — Participants will engage in an interview based in motivational interviewing
  Arms: Motivational Interview Only

SUMMARY:
The goal of the current study is to develop and test an innovative, low-burden method of post-intervention contact that is based on principles of motivational interviewing and the elicitation of change talk. Participants will be randomly assigned to an assessment only control group, a standard BMI group or a BMI + video group. Participants in the BMI and BMI + video groups will complete a semi-structured, motivational intervention. Following the intervention, participants in the BMI + video group will be asked to create a personalized video in which they speak to their future self and describe their reasons for wanting to reduce their alcohol use and their commitment to change. Doctoral level psychology graduate students will assist participants in idea generation and creation of the post-intervention video. Video group participants will then be sent their personalized videos 21 days after the baseline session, a time when motivation to reduce drinking often begins to wane. It is hypothesized that participants in the BMI + video group will rate the video exercise as helpful, encouraging, and easy to complete. It is further hypothesized that, over the 6-week intervention period, (1) participants in the BMI + video group will reduce their alcohol use more than those in the standard BMI and control groups and (2) participants in the standard BMI group will reduce their alcohol use more than those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Meets National Institute on Alcohol Abuse and Alcoholism criteria for heavy drinking
* 18 year or older
* Accessibility to internet and laptop with camera and microphone

Exclusion Criteria:

* Failure to meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Alcohol Consumption | 6 weeks post intervention
Motivation to Change Rating Scale | 6 weeks post intervention
  This outcome measure asks: On a scale of 1 to 5, how likely are you to reduce your drinking over the next week, month, and year. In this scale 1 represents not at all likely and 5 represents extremely likely.

SECONDARY OUTCOMES:
Rating Scales Assessing Satisfaction with the Intervention | 6 weeks post intervention
  This outcome measure asks participants to rate their experience with the intervention on a number of dimensions (e.g. empathic, personalized). Additionally, video participants are asked to rate the extent to which they experienced different emotions (e.g. anger, proudness) while watching their video recording. Responses range from not at all to extremely.

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States